CLINICAL TRIAL: NCT02897726
Title: A Clinical Trial to Evaluate the Pharmacokinetics and Safety of NVP-1402 in Healthy Male Subjects
Brief Title: A Study to Evaluate the Safety and Pharmacokinetics of NVP-1402
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: NVP-1402-01
Record Dates: First submitted 2016-09-01; First posted 2016-09-13 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVP-1402 (Experimental): NVP-1402 was administered once a day for 24 hours
  Interventions: Drug: NVP-1402
- NVP-1402R (Active Comparator): Active comparator was administered twice a day for 24 hours
  Interventions: Drug: NVP-1402R

INTERVENTIONS:
Drug: NVP-1402 — Oral
  Arms: NVP-1402
Drug: NVP-1402R — Oral
  Other Names: Active comparator
  Arms: NVP-1402R

SUMMARY:
The purpose of this study is to evaluate and compare the safety and pharmacokinetics of NVP-1402 and NVP-1402R in healthy male subjects.

DETAILED DESCRIPTION:
This study is designed as randomized, open-label, active-controlled and crossover assignment for evaluate and compare the safety and pharmacokinetics of NVP-1402 and NVP-1402R in healthy male subjects. The safety assessed through adverse events up to 17 days after administration. Additional variables (ECGs, laboratory test, vital signs, so on) will also be recorded and assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* No history of clinically significant medical disorder
* Capable of consent to participate in the study

Exclusion Criteria:

* History of hypersensitive reactions to study drug or other related drugs
* Any significant abnormality found during screening
* Any significant medical history
* History of alcohol abuse, smoking continuously
* History of drug abuse
* Clinically significant surgery within 4 weeks prior to administration of the study drug
* Participation in another clinical trial within 3 months prior to administration of the study drug

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of plasma: Cmax | up to 24 hours after administration
  Maximum measured concentration of the analyte in plasma
Pharmacokinetics of plasma: AUClast | up to 24 hours after administration
  Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point

SECONDARY OUTCOMES:
Pharmacokinetics of plasma: AUCinf | up to 24 hours after administration
  Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity
Pharmacokinetics of plasma: Tmax | up to 24 hours after administration
  Time from dosing to the maximum measured concentration of the analyte in plasma
Pharmacokinetics of plasma: t1/2 | up to 24 hours after administration
  Terminal half-life of the analyte in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ran Yoon, M.D.,Ph.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Navipharm, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No